CLINICAL TRIAL: NCT07270471
Title: Evaluation of Two Dermatophyte qPCR Kits on Skin and Keratinous Samples
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Anne DEBOURGOGNE, PU-PH, Central Hospital, Nancy, France
Other Study IDs: 2024-PI-081
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Dermatophytosis
MeSH Terms: conditions — Tinea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin, nail, hair
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR dermatophyte — multiplex dermatophytes PCR

SUMMARY:
Superficial fungal infections (onychomycosis, dermatophytosis, tinea, etc.) caused by dermatophytes are common in the general population, affecting 20-25% worldwide (1, 2). In our practice, the most frequently observed clinical presentation is onychomycosis, with a prevalence ranging from 2% to 16.7% (3). However, diagnosing this fungal infection is challenging due to its lack of specificity and the long culture turnaround time (up to one month). A molecular approach could overcome these two limitations.

Currently, upon sample receipt, a direct mycological examination is performed alongside culture on specific media. If culture is positive, species or genus identification is carried out. Thus, the current reference method is a positive direct examination and/or a positive dermatophyte culture. Over the past four years (2020-2023), 49.85% of samples analyzed in our laboratory were positive (direct exam ± culture).

Several PCR kits are available for molecular detection of dermatophytes in skin and keratinous samples, and initial studies report promising performance: sensitivity ranging from 78.5% to 96.5% and specificity from 89.1% to 100%.

The study aims to determine the role of molecular diagnostics in these mycodermatological conditions and to compare the performance of two commercial kits.

Primary objective:

Determine the diagnostic performance of two molecular techniques for detecting dermatophytes.

The reference technique (gold standard) will be the presence of dermatophytes established by direct fungal examination. If the direct examination is negative, fungal culture will be performed for confirmation.

Secondary objectives:

Compare the diagnostic performance of the two molecular biology kits. Compare the average turnaround time for results.

ELIGIBILITY:
Inclusion Criteria:

* Patients consulting at CHRU Nancy for suspected dermatophyte infection.

Exclusion Criteria:

* out CHRU Nancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting at CHRU Nancy for suspected dermatophyte infection.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-12-27 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
dermatophytes : yes / no and species involved | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France